CLINICAL TRIAL: NCT00498277
Title: Quantitative Diffusion and Fat Imaging of Vertebral Fractures
Brief Title: Quantitative Diffusion and Fat Imaging of the Spine
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0317
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Magnetic Resonance Imaging; Vertebral Fractures; Quantitative Diffusion; Fat Imaging; Spine
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal MRI
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — One MRI sequence done to look for relative fat, and a second extra MRI sequence done to look for the diffusion.
  Other Names: MRI

SUMMARY:
Primary Objective:

The purpose of this study is to determine whether or not combined quantitative diffusion and fat MR imaging techniques can differentiate between benign and malignant vertebral fractures.

DETAILED DESCRIPTION:
Researchers believe that they may be able to use MRI scans to tell if fractures of the bones in the spine are due to cancer. They believe this can be done by looking at MRIs of diffusion (the random motion of molecules) and fat. For benign and malignant processes, either diffusion or fat, or both of them, can be different, because the cell density (which affects diffusion) and bone marrow content (which affects fat) are expected to be different.

All patients in this study will have already been scheduled for MRI exams of the spine at UTMDACC.

You will have one extra MRI sequence done to look for relative fat, and a second extra MRI sequence done to look for the diffusion. The extra time required for the study should be less than 10 minutes, and the total imaging time should fall within a standard MRI time slot.

Available data from your medical record, including imaging data, will be used to set up guidelines and clear examples for checking spinal fractures.

This is an investigational study. A total of 48 patients will take part in the study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected vertebral compression fractures scheduled a standard of care MRI of the spine.

Exclusion Criteria:

1. Patients who are contraindicated for MRI (such as due to metal implants, cardiac pacemaker).
2. Patients who are unable to give informed consent
3. Patients who are younger than 18 years of age since the disease (osteoporosis) is not present in children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with osteoporosis that have already been scheduled for MRI exams of the spine.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
MRIs of diffusion (the random motion of molecules) and fat | One extra 10 minute MRI sequence during scheduled spine exam.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfei Ma, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org